# Study Protocol and Statistical Analysis Plan Enhancing Adolescent Substance Abuse Treatment NCT03249350

PI: Mike McCart, PhD; Oregon Social Learning Center 08/17/2017

#### SCIENTIFIC RIGOR

The proposed study will achieve robust and unbiased results via several features, including a priori hypotheses; explicit inclusion/exclusion criteria; use of well-established measures and multi-method validation of primary constructs; ensuring data collection staff are blind to treatment assignment; carefully delineated data analysis plans; power estimates; and plans for retention, missing data, and potential confounds. Biological variables (age, sex) are incorporated into the analytic plan. Study details are reported in a transparent way to support replication, and investigators expose results of all their studies to high quality peer-review procedures. **PRELIMINARY STUDIES** 

Several areas of past work culminate in this proposal: (a) mediation studies and research on the proposed direct (parent management) and indirect (behavioral regulation, peer relations) targets, (b) clinical research involving family-based CM and other EBPs, and (c) dissemination research with CM and other EBPs.

# STUDIES INVOLVING THE PROPOSED TARGETS AND MEDIATORS OF EBPS.

PARENTING AND PEER RELATIONS. The PI and Co-I's have collaborated on many studies evaluating parent management, as well as numerous studies evaluating peer relations and impacts on youth behavior (see Biosketches). In fact, the Oregon Social Learning Center (OSLC) and the PI's former institution, the Family Services Research Center (started by Co-I Henggeler), are internationally known for their contributions to studying parenting, peer relations, and high-risk youth. Thus, the team is optimal for leading this research.

NEUROCOGNITIVE PROCESSES UNDERLYING BEHAVIORAL REGULATION. For over a decade, OSLC researchers have examined the effects of stress on youths' neurocognitive functioning. Co-I Bruce has expertise in acquisition, analysis, and interpretation of data measuring risk taking and inhibitory control abilities in adolescents. 119–123 She also has expertise with neurobiological measures collected in studies of foster care and a family-based school readiness intervention for at-risk youth. 28,124–125 Of importance, results from studies employing event-related potential and event-related functional magnetic resonance imaging suggest parenting interventions can alter the neural systems underlying behavioral regulation. 28,124,126 Bruce, therefore, is well equipped to guide examination of the putative mediating effects of risk taking and inhibitory control.

MEDIATION OF EBPs. Several trials conducted by the team have produced papers examining mediators of experimental interventions. 94-95,127-128 For one manuscript, 127 McCart and Chapman co-led the complex mediation analyses. Thus, the team is equipped to accomplish the proposed work. The approach to mediation (experimental mediation) is a unique innovation, although the methods integrate standard RCT and data collection techniques with which the team has vast experience. However, to further strengthen the team's expertise, David MacKinnon, a leading experimental mediation expert, will serve as a consultant.

# CLINICAL RESEARCH INVOLVING FAMILY-BASED CM AND OTHER EBPS.

RCTs and implementation efforts involving family-based CM. As noted, family-based CM is one of several validated adolescent interventions. A variation of family-based CM developed by Azrin, Donohue et al. produced positive results in several studies. Pollowing that work, our team conducted an RCT, in collaboration with Donohue, evaluating CM combined with MST for substance abusing juvenile offenders. More recently, our team collaborated on an RCT integrating family-based CM into juvenile drug courts, as well as the aforementioned RCT comparing CM and an HIV-risk reduction protocol to TAU for delinquent youth. Study results have demonstrated significantly better outcomes for youth in CM conditions relative to controls; however, treatment effects have tended to fall in only the small to medium range.

With extensive understanding and use of Instructional Design Theory (advocated by educational researchers 132-134), the investigative team has focused on developing family-based CM suited for training and implementation in real world settings. In fact, McCart and Sheidow started a clinic at their prior institution that utilized Master's level practitioners to deliver CM to the local community and have developed a similar capacity at their current institution's clinic. Aside from studying its effectiveness, the team has extensive knowledge on implementation of CM, a requisite for the proposed study. Specifically, the team has experience with: (a) the range and magnitude of incentives for youth, (b) developing reward systems that leverage the empirically demonstrated impact of escalating reinforcers and rapid resets (a "leveled" system), 135-136 and (c) blending immediate reinforcers (immediate access to most valued privileges) with a token economy system (accruing points to purchase from individualized and varied reward/privilege menus). With this experience delivering family-based CM in clinical research and real-world practice settings, the team is primed for the proposed trial.

RCTs AND IMPLEMENTATION EFFORTS INVOLVING OTHER EBPs. The PI and Co-l's also have conducted numerous RCTs on interventions other than family-based CM. For example, McCart, Sheidow, and Chapman are collaborating on RCTs of interventions for victims of child sexual assault (R01DA031285) and youth with comorbid mental health and substance use problems (R01DA025616). Further, Henggeler has 3+ decades of experience conducting RCTs on MST and other family-based youth treatments (e.g., several RCTs with violent juvenile offenders, 137-139 two with substance abusing juvenile offenders, and one for youth with serious emotional disturbance 140). Similarly, Chamberlain conducted several RCTs of TFCO for antisocial youth. 141-142

Of note, these trials all included close collaboration with community agencies, random assignment, evaluation of multiple outcomes, and minimal exclusion criteria to enhance external validity. These trials also

had diverse samples (e.g., <u>up to 32% Latino, 81% African American, 12% Native American</u>) and high recruitment rates (see details in *Recruitment and Retention Rates* section). Thus, the investigators are skilled at implementing intervention protocols, recruiting diverse youth and families into clinical research, executing data collection protocols, and performing advanced data analyses to answer research questions.

# DISSEMINATION RESEARCH WITH FAMILY-BASED CM AND OTHER EBPS.

The study also is supported by our work transporting CM and other EBPs to community settings. The investigators completed several NIDA-funded studies examining CM transport to the public sector including: a study of quality assurance on CM fidelity among providers in Connecticut<sup>117</sup> and a replication in Norway;<sup>143</sup> a 44-site Statewide Study on training 432 therapists in CM and examining their adoption;<sup>35–36</sup> and a CM Training Study evaluating relative effectiveness of different training methods among 100+ public sector therapists.<sup>144</sup> Findings from the Statewide Study indicated strong interest, with 80% attending a workshop and 58% adopting CM. Adoption was related to individual characteristics and attitudes toward EBPs; negative attitudes toward CM was not a barrier cited. Other investigators have examined transportability of CM to community settings and found high adoption rates.<sup>145-147</sup> The team also has researched transportability of other EBPs. For example, Sheidow and Chapman collaborated with Sonja Schoenwald on a 45-site MST transportability study, which indicated (a) a complex intervention can be transported to community-based therapists, (b) fidelity predicts outcomes, and (c) clinician and organizational factors affect fidelity and outcomes.<sup>148</sup>

**CONCLUSION.** The team has extensive experience evaluating and transporting EBPs. Our research suggests that while family-based CM is a well-validated EBP for adolescent SUD, its effects, like other adolescent SUD EBPs, are modest. Thus, this study will use an experimental mediation approach to identify mediating processes in treatment, with the ultimate aim of improving SUD treatment effectiveness. Backed by our experience conducting mediation and clinical studies, this study is poised to produce crosscutting implications for improving youth SUD treatments. Given the clear need to enhance effectiveness and durability of existing interventions, such work could have a dramatic impact on outcomes and services for youth.

# DESIGN TIMELINE AND OVERVIEW

Data will be from a Ionaitudinal twoarmed parallel group design with 172 youth randomized to CM vs. CM+. In-person assessments will be at baseline, 2-, 4-, 6-, 9-, and 12-months postbaseline. Phone assessments will be at 1-, 3-, 5-, 7-, and 8months post-baseline.



# STUDY SITES

The proposed study will be conducted with the OSLC outpatient clinic and Centro Latino Americano (CLA). Both are Medicaid-approved, HIPAA-compliant clinics employing Certified Alcohol and Drug Counselors (CADC) to deliver treatment services. While the two clinics serve all Lane County residents, CLA clients are predominantly Latino. As noted in the *Introduction*, adding CLA as a second site for this trial allows for oversampling of Latino youth, permitting an examination of differential mediation effects by ethnicity (see *Data Analysis*). Importantly, OSLC scientists regularly collaborate with OSLC clinic staff on intervention trials involving methods consistent with the proposed study. Similarly, OSLC scientists have a long history of collaborating with CLA on research and implementation projects. 149-150 Thus, the sites are optimal for ensuring adequate recruitment numbers, protocol fidelity, and successful completion of study procedures.

The trial will involve 6 CADCs across the sites; 3 CADCs (2 from OSLC and 1 from CLA) will be randomly selected to deliver CM+ and the other 3 CADCs (2 from OSLC and 1 from CLA) will deliver standard family-based CM. Based on our experience with RCTs, we anticipate turnover and have planned for as-needed recruitment of new CADCs and case re-assignment to ensure cases remain within condition. To ensure high fidelity and reduce confounding variables (e.g., access, insurance), the study will pay for treatment in both conditions, and investigators will train and closely monitor CADC staff.

Adolescents presenting to OSLC and CLA for SUD treatment during Study Months 7-42 will be screened, and those meeting inclusion criteria will be offered the opportunity to participate pending available slots. Power calculations (presented subsequently) indicate an optimal sample size of 172. Given case flow at the clinics, and our desire to oversample Latino families, we anticipate achieving the required sample size in 3 years. Specifically, CLA treats 23 adolescents with SUD per year on average, and all of these will be approached to participate in

the trial. Assuming an 80% recruitment rate (see subsequent rationale for this rate), we expect to recruit 55 families from CLA across the 3 years. OSLC serves just over 100 cases/year on average, so case flow will provide more than enough families to recruit the remainder of the sample (49/year x 3 years = 117). Based on information from OSLC and CLA, the following demographic characteristics are expected for youth recruited across both clinics: average age = 15 years (range = 12-17 years); 84% White, 13% African American, 2% American Indian/Alaska Native, 1% Asian; 35% Latino (of any race); and 30% female.

#### **PARTICIPANTS**

Participants will include 172 youth and their primary parent/guardian. Inclusion criteria for the youth are: 1) age 12-17 years; 2) presence of current SUD; and 3) availability of a parent/guardian willing to participate. Exclusion criteria are: 1) actively psychotic, suicidal, or homicidal; and 2) PDD or mental retardation. To increase external validity, youth will be included regardless of co-morbid mental health or physical difficulties.

# RESEARCH SCREENING, RECRUITMENT, AND RETENTION

**INITIAL SCREENING.** All cases presenting to the OSLC and CLA clinics meet initially with an intake worker to determine appropriateness for an outpatient level of care. The intake worker will make a preliminary determination regarding study eligibility and refer them and their parents to Project Assessors.

**STUDY RECRUITMENT AND SCREENING.** Assessors will meet with youth and parents at a time and place convenient to the family (clinic, family's home, private community location) to obtain parental consent/youth assent. Protections will be assured, including IRB approval and a federal Certificate of Confidentiality. After this, SUD will be confirmed via the Global Appraisal of Individual Needs-Initial, Lite (GAIN-I, Lite), 151-154 a diagnostic interview aligned with the DSM-5. If lacking a SUD, youth and parents will each be provided \$10 gift cards. If SUD is present, a 2-hour baseline interview will be conducted and subsequent interviews scheduled.

**RECRUITMENT AND RETENTION RATES.** In over 15 years conducting treatment research with families, we have achieved recruitment rates ranging from 85-100% and retention rates exceeding 90% for 12-month follow-ups. 34,55,107 The research team has been very successful at recruiting and retaining participants from challenging populations, and the majority of these studies were conducted in real world (rather than research) clinics where youth/families could receive treatment without consenting to research. We will replicate our successful recruitment and retention strategies in this trial. First, to establish collaborative relations with families, assessments are scheduled at their convenience, contacts are as friendly as possible, and families are reimbursed for their time. Second, direct contact helps maintain the cohort, with families contacted regularly during their 12 months of study participation. At each contact, families are asked if they plan to move and for up to 4 phone numbers and email addresses of best friends, relatives, and schools/places of employment. Third, we obtain consent to use technology such as text messaging and Facebook (using private messaging functions). When participants cannot be located, Assessors track them using the various contacts, other Internet resources (e.g., reverse look-up), and post office forwarding. Fourth, the same Assessor follows participants over time to encourage rapport. Fifth, contacts are defined as confidential and independent of treatment. Reasons for missed interviews will be recorded to assess impact on proposed methods.

# **RANDOMIZATION TO CONDITIONS**

An adaptive urn randomization procedure, <sup>155-158</sup> implemented using the Microsoft Access application gRand, will balance potential confounding variables among participants randomized to each condition and also will manage condition sizes. This method is recommended for trials of SUD treatments. <sup>155</sup> Based on the population and outcomes of interest, factors on which the urn will operate are youth age, sex, baseline substance use severity, and a weighted percentage schedule for condition balance. The urn will minimize variability in these pre-treatment variables across the two conditions. To keep Assessors blind to condition, the Assessment Coordinator will conduct the randomization procedure immediately following a family's baseline assessment and will convey results directly to parents. The Coordinator also will inform the clinic intake worker of the randomization result so the family can be assigned to a CADC in the correct condition: CM+ or CM only.

# **DATA COLLECTION PROTOCOL**

Assessors will meet with youth and parents for (1) a 2-hour, in-person baseline interview, (2) in-person, 1.5-hour follow-up assessments at 2-, 4-, 6-, 9-, and 12-months post baseline, and (3) 30-minute phone interviews at 1-, 3-, 5-, 7-, and 8-months. If youth and parent have to be assessed at different sessions, they will be scheduled within one week of each other. This schedule provides frequent measurement of constructs during active treatment (both CM+ and family-based CM are expected to last 5-6 months on average), while also providing a longer view on durability of change than is typical in adolescent SUD treatment research.<sup>19</sup>

To compensate for their time, families are paid \$50 for baseline and \$40 for each in-person follow-up assessment. Families will be paid \$10 for each brief telephone assessment (maximum total compensation = \$300). Based on our experience, 1.5- to 2-hour assessments rarely present a significant response burden, but Assessors are trained to use breaks with snacks and to attenuate circumstances that threaten validity of assessments. Participant protections are detailed in the Human Subjects Protocol and include IRB approval.

# **M**EASURES

Multiple methods or perspectives will enhance construct validity. Consistent with intention-to-treat principles,

data from all time points will be collected even if families drop out of treatment.

#### Table 2. Research Instruments

# Descriptive Variables [Baseline only]

Structured Adolescent Interview<sup>159</sup> for demographics and to supply relevant data for the urn randomization.

# Ultimate Outcomes [Months 0, 2, 4, 6, 9, & 12]

#### SUBSTANCE USE:

**Urine samples** collected by researchers from youth; lab testing for THC, synthetic THC, amphetamines, opiates, PCP, cocaine, and alcohol metabolites (EtG/EtS); selected lab's testing procedures are of high scientific quality.

**GAIN**<sup>151-154</sup> scales measuring self-reported youth substance use and substance-related problems; 16-item substance abuse index/substance dependence, substance problem scales assessing DSM-5 criteria for substance use disorders and lower severity symptoms, recovery environment risk and social risk subscales that predict substance-related problems in youth with substance abuse, and the substance frequency scale assessing substance use for past 90 days; GAIN scales have good reliabilities and sensitivity to change, and are highly associated with results from Form-90 and urine testing. <sup>160-161</sup>

**EXTERNALIZING BEHAVIOR:** Externalizing subscale of parent-completed **Child Behavioral Checklist** and corresponding subscale of **Youth Self Report**; <sup>162</sup> scales provide valid measures of youth externalizing behavior from multiple perspectives. <sup>163</sup>

# Direct Target [Months 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, & 12]

# **PARENT MANAGEMENT:**

**Alabama Parenting Questionnaire (APQ)**<sup>164</sup> administered to youth and parents, measuring monitoring/supervision, positive parenting (social/tangible reinforcement), and consistent discipline (removal of privileges); scales have been used to document treatment outcomes and distinguish families of youth with and without behavior problems; <sup>164</sup> scales have established reliability and validity; <sup>165</sup> an additional rules and expectations subscale added to the APQ assesses enforcement of household rules.

**CM Adherence Measure (CAM)** developed using Rasch methods and validated across several studies with substance using adolescents;<sup>37,166-167</sup> subscales measure cognitive behavioral (antecedent-behavior-consequence assessments, self-management planning) and behavioral (drug screening, contingency contracting) techniques used within family-based CM. Originally, this tool was designed for families to rate their therapist's delivery of CM in session. However, as noted previously, a central feature of CM is to train parents to continue implementing CM at home. Thus, for this study, parent and youth CAM reports will be obtained to assess parents' implementation of CM both between the sessions and after treatment has ended.

# Indirect Targets [Months 0, 2, 4, 6, 9, & 12]

**PEER RELATIONS: Pittsburgh Youth Study**<sup>111</sup> scales with strong reliability and validity;<sup>168</sup> youth-reported peer delinquency scale and drug activity scale measuring proportion of youths' friends who engage in antisocial behaviors per youth report, youth-reported conventional activities of peers scale measuring proportion of friends who engage in prosocial activities, and bad friends scale assessing youth contact with peers disapproved of by parents per youth and parent report.

# **BEHAVIORAL REGULATION - RISK TAKING:**

**Behavioral Inhibition System (BIS) and Behavioral Activation System (BAS) Scales** completed by youth and parents; <sup>169–170</sup> BIS is sensitive to signals of punishment and non-reward; BAS is sensitive to signals of reward; BAS includes three subscales: drive (persistent pursuit of desired goals), fun seeking (spontaneous desire for new rewards), and reward responsiveness (positive responses to the anticipation of rewards); scales have satisfactory reliability and validity. <sup>169–170</sup>

**Balloon Analogue Risk Task - Youth** assesses risk-taking propensity. 81,171 Adolescents earn points every time they pump to inflate a computer-generated balloon, a computer algorithm randomly determines the number of pumps that will cause the balloon to pop, and the adolescents lose points if the balloon pops. An index of risk taking is calculated by averaging the number of pumps for balloons that did not explode. 81 The task has good internal consistency and convergent validity. 81

# BEHAVIORAL REGULATION - INHIBITORY CONTROL:

**Early Adolescent Temperament Questionnaire–Revised**<sup>172–173</sup> completed by youth and parents; scales include inhibitory control and higher-order factors: effortful control, negative affect, affiliativeness, extraversion; good internal consistency.<sup>173</sup>

**Go/No Go Task** of inhibitory control; youth selectively respond to target stimuli and inhibit responses to equally salient, non-target stimuli. 121,174 Consists of 252 trials: a letter is presented for 500-ms with a fixed, 1,500-ms interstimulus interval. Youth is instructed to press button as quickly as possible for every letter (go stimuli) except X (no go stimuli); 75% "go" trials and 25% "no go" trials; activates dorsolateral prefrontal cortex, ventral prefrontal cortex, and anterior cingulate cortex. 174 Consistent with prior research, 175–176 we will compute an index of inhibitory control: subtract percent correct on highly interfering stimuli ("no go" trials) from percent correct on minimally interfering stimuli ("go" trials). Lower scores indicate better inhibitory control.

#### TREATMENT CONDITIONS

**FAMILY-BASED CM**. Family-based CM is rooted in behavioral and cognitive behavioral theories and is designed for delivery in outpatient clinic settings (weekly 50-60 minute sessions). Treatment duration is criterion-based, determined by achievement of substance use goals, but the protocol is typically 5-6 months (20-24 sessions). CM has strong empirical support in the adult SUD treatment literature, <sup>177</sup> and family-based CM has also proven efficacious for youth SUD. <sup>13,178</sup> Moreover, its relative simplicity and low cost <sup>179</sup> makes family-based CM highly amenable to adoption. The protocol components are listed in Table 3.

# Table 3. Family-Based CM Components

**Clinical assessment.** A semi-structured interview conducted separately with the youth and parent gathers type, frequency, quantity, and administration route of drug use; and data on treatment, medical, and educational history.

Introducing CM. CM is introduced to the youth and parent, and the therapist begins to engage them both in treatment.

**Antecedent-behavior-consequence (ABC) assessment.** ABC assessments of the youth's substance use are conducted in collaboration with the youth and parent (similar to functional analyses), in which they are asked to identify environmental, cognitive, and affective triggers (i.e., antecedents) for recent episodes of use or abstinence and to reflect on both the positive and negative consequences of that use/abstinence. ABC assessments are completed in each session, but parents and youth also are trained to complete these together as homework following each drug test completed at home (see below).

**Self-management planning.** The triggers identified in ABC assessments are targeted via self-management plans developed by the therapist, youth, and parent. Plans commonly fall into three categories: (a) avoiding triggers (e.g., avoiding certain peers, decreasing time spent in places/with people that trigger use while increasing time spent in places/with people that trigger abstinence), (b) rearranging environment (e.g., purging items associated with drug use), and (c) developing effective drug refusal skills for unavoidable triggers such as peer pressure. Once a list is generated, the therapist helps the youth and parent weigh the potential costs, benefits, and difficulty level of each strategy so they can choose the best plan.

**Drug testing and contingency contracting.** Concurrent with developing self-management plans, parents are taught to conduct random urine drug screens and breath scans at home. Screens also are conducted at every scheduled treatment session. Finally, the therapist and parent arrange for periodic random clinic visits to conduct screens. The therapist, youth, and parent create a contingency contract that specifies consequences based on the results of the screens.

The contingency contract follows a well-specified protocol for behavior plans. First, the therapist, youth, and parent generate a menu of rewards that can effectively compete with the youth's substance use. The therapist ensures there is a balance between natural incentives parents can provide (e.g., cell phone access; later curfew) and items to be purchased with gift cards (i.e., therapists have access to \$250/youth for gift cards). To assist therapists and parents in identifying rewards with the best odds of competing with substance use, rewards are rank ordered by the youth based on preference. From this reward menu, the youth and parent choose the youth's "most valued privilege" (MVP), which is almost always a natural incentive a parent can provide regularly. Remaining menu items are assigned point values by the parent and therapist, usually 1 point ≈ \$1. Once the menu is finalized, a point-and-level system is implemented and the youth receives a 50-point starting balance. The youth earns or loses MVP access from the parent depending on each drug screen result. During the first month (Level I of the contract), youth keep their points if they have negative drug screens, but lose 12 points for each week they test positive. Regardless of screen results, youth cannot redeem their points in this period. From the fifth week on (Level II of the contract), negative screens result in youth being able to earn additional points and also to use their points to "purchase" items on the reward menu. To provide a greater incentive (i.e., escalating reinforcer), the number of points youth can earn each week starts at 12 and then increases to 24 after eight consecutive weeks of negative drug screens (Level III of the contract; rapid reset is also used). When making a purchase, youth may use as many points as they would like from their balance. Rewards are provided as immediately as possible, consistent with behavioral principles. If a youth has a positive screen from the fifth week on, the youth does not earn points and cannot make a "purchase" until the next negative screen. As treatment progresses, emphasis shifts to using natural incentives provided by parents to sustain abstinence and also expansion of the behavior plan to include any other behaviors the parent wants to target.

**CM+ TO ENHANCE PARENT MANAGEMENT.** As discussed, although family-based CM involves parent participation, evidence indicates it does not yield reliable improvements in parent management skills. Consistent with the enhancement manipulation-of-mediator design, an approach was chosen to target the putative parenting mediator more intensely in CM. In selecting the approach, the following criteria had to be met. It needed to be: (a) powerful enough to generate meaningful changes in parenting, (b) conceptually consistent with CM, and (c) feasible for delivery in outpatient settings. Various approaches were considered, and the well-validated behavioral assessment and teaching system from PMTO² was ultimately chosen. This system was selected for three reasons. First, PMTO is supported by five decades of efficacy, effectiveness, and implementation research, and it is the leading parent training intervention for youth. <sup>180</sup> Indeed, evaluations of PMTO with child and adolescent samples demonstrate it produces substantial reductions in youth externalizing behavior. <sup>181</sup> Second, and of central importance to the present proposal, mediation studies indicate that the behavioral assessment and teaching system in PMTO produces improvements in parent management skills, and those improved skills largely account for PMTO's effects on youth outcomes. <sup>180</sup> In fact, of all parenting interventions, PMTO has the most support for improved parenting as the key mechanism of action. <sup>180</sup> Third, PMTO has been extensively tested and validated for use with diverse samples, including Latino families. <sup>182</sup>

PMTO was developed and validated by OSLC scientists in the 1970s, and this EBP is currently being implemented in over 100 national and international sites.<sup>2</sup> The model is comprised of a *behavioral assessment and teaching system* as well as *clinical content*. In PMTO, the *clinical content* is typically behavioral concepts focused on externalizing problems, but can be tailored by subpopulation. Thus, CM strategies (detailed above) can be the clinical content. PMTO's *behavioral assessment and teaching system* was developed as the specific therapeutic processes used to deliver the clinical content and the system is viewed as critical to achieving PMTO's meaningful change in parenting.<sup>182</sup> In essence, the system involves "parallel processes" in that it employs behavioral principles, the same behavioral principles employed to change the child's behavior, to facilitate parents' active learning and rapid skill acquisition. As such, the PMTO *behavioral assessment and teaching system* can be seamlessly adopted by other conceptually consistent interventions. Indeed, Co-l Chamberlain has incorporated this system into both TFCO<sup>183</sup> and KEEP.<sup>184</sup> Similarly, with oversight from

Chamberlain, the CM+ protocol will add the *behavioral assessment and teaching system* from PMTO to standard CM to enhance parent's skill acquisition more intensely (see Table 4).

# Table 4. PMTO Behavioral Assessment and Teaching System Incorporated Into CM

This system uses three fundamental **Processes** (listed below) to bring about changes in parenting. These processes are interdependent therapeutic operations, <sup>185</sup> forming the fundamental skills a therapist employs. The basis for these processes is to address a youth's behavior problems using methods based on behavioral principles to change the parent's behaviors. These processes are the therapeutic skills used to deliver clinical content (i.e., to assess and teach parent management) and are based on principles of *behavioral chaining*, *shaping*, *fading*, *generalization*, *immediacy*, *reinforcement*, *differentiation*, *cueing*, and *modeling*.

Parent Daily Report (PDR1). The PDR procedures entail highly structured phone calls to the parent. Although the PDR typically includes daily phone calls, we believe it would be more feasible and prevent potential barriers if phone calls were conducted every other day (i.e., approximately twice between sessions). Calls are pre-arranged to occur at convenient times for the parent. Parents are oriented to PDR procedures so they are prepared for how the structured call will be conducted. First, the therapist ensures the parent can speak confidentially (ensure privacy). The therapist then asks a series of brief questions assessing occurrence/nonoccurrence during the past 48 hours of specific adolescent behaviors (e.g., adherence to rules, substance use confirmed by urine drug screens), parental responses to those behaviors (e.g., reinforcement, limit setting, supervision), and the youth's reactions to the parental response. The therapist then offers guidance and feedback (cueing) to parents on effective parent management techniques. These include breaking complex parenting behaviors into smaller steps (behavioral chaining) and providing positive feedback (reinforcement) in proximity to specific parent management accomplishments (immediacy). Rather than focus on all parenting behaviors, the parenting behaviors (including smaller steps in the behavioral chain) are rank ordered by the therapist prior to the calls so the therapist can focus on a single parenting behavior for each phone call (based upon the combination of prioritization and occurrence/nonoccurrence of behaviors: fading and shaping of parent management skills). The therapist also graphs parenting behaviors based on PDR data collected in each call; the graph is used to illustrate progress during in-person treatment sessions. Research indicates that when implemented with other behavioral interventions, the PDR is highly feasible and has good utility for improving parent management skills. 186-189 Also of importance, the PDR is easy to implement and fits within the practice parameters of outpatient therapists (contacting and guiding parents in specific skills related to the youth's treatment).

**3-D Role-Play.** Therapists are trained in this method to help parents develop and refine the use of parenting skills. Although role-play is not a new technique, OSLC scientists developed the 3-D method in collaboration with Salvador Minuchin (developer of Structural Family Therapy) to enhance its capacity as a teaching tool. <sup>190</sup> The therapist first meets individually with the parent to Demonstrate an ineffective response to a problematic youth behavior, such as lecturing. Next, the therapist models a more effective strategy, such as swiftly implementing a consequence in a calm voice, to Differentiate it from the ineffective approach (differentiation and modeling). Finally, the therapist and parent Debrief to consider positive and negative consequences of the ineffective and effective strategies. Reflective questioning during debriefing increases parents' awareness of how their verbal and nonverbal behaviors influence interactions with their youth (cueing). For example, therapists might ask, "What did I do to make you want to cooperate? How was my tone of voice?" Such 3-D role-plays are used in every session to facilitate step-by-step learning of complex skills (behavioral chaining), with each step representing a small change that contributes to successful implementation (shaping). Once a parent becomes proficient with a skill, s/he is assigned homework to try it in real-life situations (generalization). After opportunities for testing, skills are revisited during sessions and PDR calls and refined for future application (generalization).

Anti-Coercive Problem-Solving. Teaching a parent to change his/her parent management skills requires instruction. A collaborative problem-solving approach was developed based on research indicating that parental resistance to this instruction (a high base rate phenomenon in parenting interventions) can be exacerbated or abated by therapist responses. 191 Instead of straightforward instruction, therapists are trained to demonstrate (modeling) problem-solving steps (identifying goal statements, brainstorming options, identifying manageable steps to achieve goals) and to use those steps as clinical skills to prevent or manage resistance. Problemsolving begins in the first session as therapists help parents articulate goals for their child's treatment. Parents learn to break goals into small achievable steps (behavioral chaining), and progress is tracked and praised at every session (shaping and reinforcement). Brainstorming becomes a strategy to engage parents and manage resistance. For example, if parents express doubt about their ability to complete a task, such as withholding an MVP if their youth tests positive for drugs, the therapist avoids engaging in a coercive interchange and collaboratively brainstorms solutions instead. Parents might decide to solicit assistance from another adult family member in withholding the MVP or decide to change the MVP to an item they can more confidently withhold (shaping). Thus, active problem-solving is always emphasized. Further, because behavior plans rarely work perfectly on first attempts, therapists provide strategic warnings to help parents anticipate that their plans might need revision (cueing). This approach increases parents' comfort in reporting challenges with implementing a behavior plan. Whenever this occurs, the therapist emphasizes positive aspects of the parent's effort at implementing the plan (shaping) while identifying areas for refinement, helping the parent create a new plan, and rehearsing new skills via role-play practice, as needed.

Of importance, our team's decades of clinical experience with the PMTO behavioral assessment and teaching system supports feasibility of implementing it as part of CM+. Indeed, OSLC staff implement the PDR each day with hundreds of foster parents participating in TFCO throughout the U.S., with PDR completion rates ranging from 70-100%. In addition, the behavioral assessment and teaching system is actively being utilized in programs at the OSLC outpatient clinic. As an example, for over seven years, OSLC therapists have served a population of parents referred by child welfare due to serious substance abuse and neglect of their children. As a central component of that outpatient treatment, therapists administer PDRs to parents every other day (consistent with the proposed CM+ schedule) and use the PMTO role-play and problem-solving strategies to enhance parents' delivery of effective parent management skills. OSLC staff have achieved a PDR collection

rate of 79% and a treatment completion rate of 81% with these high-risk substance-abusing parents, highlighting the feasibility of delivering these strategies in an outpatient clinic.

**ACHIEVING AND ASSESSING FIDELITY.** Treatment fidelity is essential for internal validity (ensuring standard family-based CM and CM+ are implemented as intended and differ from one another only with regard to the experimental enhancement). Thus, strong treatment fidelity is critical to establishing effectiveness, and a well-developed protocol will be used for training and ongoing quality assurance. Specifically, therapists in both conditions will receive training and ongoing quality assurance from McCart and Sheidow. The training protocol follows that used in our other family-based CM research and large-scale transport of CM to community-based practitioners. <sup>35–36</sup> An initial 3-day workshop orients clinicians to program philosophy and all intervention methods. Clinical supervision further supports therapists' implementation, modeled on a structured CM supervisory manual. <sup>192</sup> Following workshop training, clinicians practice treatment delivery to families and have individual supervision weekly to review progress and problem-solve barriers. As high fidelity becomes consistent, weekly phone coaching is provided, focusing on fidelity and solutions to difficult clinical problems. Bi-annual booster trainings are conducted on difficulties in fidelity or achieving clinical outcomes.

Further, therapist implementation of interventions will be measured from the perspective of the youth, parent, and therapists (via self-report) and McCart and Sheidow (via coding of taped treatment sessions and PDR calls). As noted, the 34-item CM Adherence Measure (CAM) was developed using Rasch methods and validated across several studies. 166 CAM subscales measure the cognitive behavioral and behavioral interventions used in CM. Using the same format, items will be created to capture PMTO enhancements in CM+. Using standard procedures employed in our other CM studies, parents and youth will complete CAMs monthly by phone (for duration of treatment) to report on therapist's CM implementation. Investigators will monitor CAMs monthly for ongoing quality assurance and as-needed therapist remediation. In addition, a more immediate fidelity assessment and remediation mechanism will be therapists completing CAMs after each session and phone call to report on their own behavior. Further, therapists will record all treatment sessions and phone calls. McCart and Sheidow will complete observational ratings 167,193 on randomly selected (20%) treatment sessions and (20%) calls. Employing procedures used successfully in Azrin et al. 129 to monitor and improve fidelity, ratings will be compared to therapist report from the same session/call. Inconsistencies between therapist self-report and observational ratings will trigger remediation training and more intensive supervision. Session/call notes and reports also will be evaluated weekly to ensure fidelity across conditions.

**BALANCING THERAPIST CHARACTERISTICS ACROSS CONDITIONS.** We anticipate that 3 therapists will deliver CM, and 3 different therapists will deliver CM+. Prior to beginning youth recruitment, therapists will be randomized to provide services in either the CM or CM+ conditions. To minimize bias, therapists will be balanced as much as possible, given the small sample, by age, sex, race, and years of experience.

ADDRESSING RISK OF CONTAMINATION. Both treatment arms are conducted within a clinic, raising concerns of potential contamination between therapists in the same clinic. Nevertheless, based on our experience conducting RCTs, we view this risk as low. Indeed, CM and the PMTO enhancements are highly structured, requiring initial training and supervision specific to identifying barriers to treatment fidelity. Across numerous trials for similar interventions, we have found therapist fidelity varies. 194-196 More generally, research indicates even experienced therapists revert to prior/usual practice in the absence of formal structures such as ongoing supervision. 36 Thus, it is unlikely that a standard CM therapist who inadvertently hears about PMTO strategies would be able to implement them with fidelity, especially in the absence of training or access to materials and supervision. Nevertheless, contamination risk will be mitigated in several ways. First, therapists deliver treatment in only 1 condition. Second, only therapists within the condition have access to resources to facilitate implementation. Third, clinical supervision is conducted individually, not in groups. Fourth, therapists formally agree not to discuss CM and CM+, except with therapists in the same condition. Fifth, as described, we measure implementation in both conditions, allowing close monitoring for potential contamination during the trial. Any evidence of contamination will be addressed immediately with therapists.

# **DATA ANALYSIS STRATEGY**

The design leads to 11 measurements of the direct target (parent management; level-1), 6 measurements of indirect targets (behavioral regulation, peer relations; level-1), and 6 measurements of ultimate outcomes (substance use, externalizing behavior; level-1) nested within 172 youth/parents (level-2). Analyses will use latent growth curve formulations of mixed-effects regression models. These highly flexible models accommodate variability in number and spacing of measurements, discrete (i.e., urine drug screens [UDS]) and continuous (i.e., parent management, behavioral regulation, peer relations, GAIN scores, externalizing behavior) outcomes, and separate patterns of change for distinct phases (i.e., during- and post-treatment).

**EXPERIMENTAL MEDIATION AND CAUSAL INFERENCE.** The experimental mediation design emphasizes evidence supporting causal inferences, and there are important conceptual and statistical considerations. As reviewed by MacKinnon, <sup>199</sup> by randomizing youth/parents, the effect of CM+ on parent management is a causal estimate. However, the effect of parent management on drug use and externalizing behavior is not straightforwardly causal, it is potentially influenced by unmeasured confounding variables. Following MacKinnon's

recommendations, and to support causal inferences, this is addressed in 3 ways. First, the enhancement design directly targets the mediator—increasing probability of a causal effect between mediator and outcome. Second, longitudinal measurements of the mediator and outcomes address temporal sequencing—demonstrating that mediator effects occur before outcome effects. Third, supplemental models evaluate confounding variables—providing evidence that mediator effects are not due to confounders.

**MODEL FORMULATION**. The underlying model is a mixed-effects latent growth curve model with repeated measurements (level-1) nested within youth/parents (level-2), implemented in Mplus (v7.31;<sup>197</sup>). As reviewed by MacKinnon,<sup>200</sup> there are several options for modeling longitudinal mediation. Flexibility of growth models for targeting phase-specific change<sup>201</sup> are leveraged and combined with parallel process models for mediation.<sup>202</sup> In a single model, there are separate change estimates for during- and post-treatment phases, directly addressing temporal sequencing of mediators and outcomes. The UDS outcome is modeled using a Bernoulli distribution, and remaining ultimate outcomes, direct targets, and indirect targets are modeled with normal distributions. Time terms are computed using assessment dates.<sup>203</sup> Treatment condition is a youth/parent-level predictor (level-2; CM = 0, CM+ = 1), and cross-level interactions are specified between condition and level-1 growth and phase terms. Models, as indicated, control for age, sex, race, ethnicity, SES, and treatment history. Likewise, preliminary models test, and control, for differences in outcomes across therapists and clinics. Follow-up models determine whether individual paths and mediated effects differ for males and females.

**STATISTICAL TEST FOR MEDIATION**. The test for mediation is based on the product of coefficients (i.e.,  $\alpha\beta$ ) with asymmetric bootstrapped *SE*s and 95% CIs for the product.<sup>204</sup> This test requires estimation of two parameters and their *SE*s, where, for example,  $\alpha$  is the effect of CM+ on parent management and  $\beta$  is the effect of parent management on substance use and externalizing behavior. Parameters are obtained from Mplus and supplied to PRODCLIN<sup>205</sup> for the asymmetric boostrapped *SE*s and CIs. This approach offers enhanced statistical power<sup>206</sup> and applies both to multilevel data<sup>207</sup> and longitudinal mediation.<sup>200</sup>

# **EVALUATION OF SPECIFIC AIMS**

AIM 1: DETERMINE WHETHER PARENT MANAGEMENT SKILLS (DIRECT TARGET) MEDIATE THE EFFECT OF TREATMENT ON YOUTH SUBSTANCE USE & BEHAVIOR PROBLEMS (ULTIMATE OUTCOMES). The test for mediation requires the coefficient and SE for CM+'s effect on parenting (a-path) and parent management's effect (controlling for treatment) on substance use and externalizing behavior (b-path). Of note, a preliminary model evaluates the direct effect of CM+ on substance use and externalizing behavior (c-path), though as noted by MacKinnon, <sup>199</sup> mediation should be tested regardless of this path's significance.

**a-path**. This model is specified with 11 repeated measurements of parenting as the outcome. To address temporal sequencing, the model estimates separate change rates for during- and post-treatment phases. This is tailored to each youth's course of treatment using coding strategies for discontinuous (piecewise) change (see Singer and Willett<sup>201</sup>). Changes during treatment phase are modeled with linear and quadratic terms for number of months since baseline. A dichotomous phase indicator differentiates post- and during-treatment measurements, and post-treatment change is modeled as linear and quadratic terms for number of months since treatment end. This provides three estimates: during-treatment slope (estimate of interest for mediation test), overall shift in parenting levels from during- to post-treatment, and post-treatment slope.

**b-path**. This model is more complex, simultaneously evaluating the mediator and outcome processes. To obtain this coefficient, the a-path is modeled along with the outcome model (c-path; testing for differences between CM+ and CM on substance use and externalizing behavior). With fewer outcome measurements, the model includes a during-treatment slope term and indicators to differentiate 9- and 12-month assessments, providing three estimates: during-treatment slope, change at 9 months, and change at 12 months. To obtain the b-path coefficient, a regression is specified with *during-treatment mediator slope* as a predictor of *outcome at 9 and 12 months*. This provides a targeted test of mediation, with during-treatment change in the mediator as a predictor of post-treatment outcomes.

**Ethnicity effects**. In close consultation with project consultant MacKinnon, and to address potential for differential effects across project clinics, formal moderated mediation tests can be performed.<sup>208-209</sup> These tests determine whether observed mediation effects differ for Latino and non-Latino youth/parents. Sample size means that results are hypothesis-generating and thus will focus on estimation of confidence intervals. The same approach will be used to evaluate moderated mediation for ethnicity in Aims 2 and 3.

**Confounding variables**. Although randomization, the enhancement mediation design, and models addressing temporal sequencing increase the likelihood of valid causal inferences for mediation, a remaining assumption is that there are no unmeasured confounding variables for the mediator's effect. Cox et al.<sup>210</sup> recommends sensitivity analyses for confounder bias be used. First, VanderWeele's<sup>211</sup> formulas identify youth/parents with the same value on the mediator but different values on the outcome, as well as youth/parents with the same value on the mediator across both CM and CM+ groups. Second, residuals from the models just detailed should be uncorrelated, and Mplus code from Imai et al.<sup>212</sup> is used to determine whether the mediated effect differs based on unmeasured pre-treatment variables. Third, Mauro's<sup>213</sup> correlational method evaluates the sources of error variance from the mediation model, determining how large the effect of an omitted variable

would need to be to negate the mediated effect.

AIM 2: DETERMINE WHETHER PARENT MANAGEMENT SKILLS (DIRECT TARGET) MEDIATE THE EFFECT OF TREATMENT ON YOUTH BEHAVIORAL REGULATION & DEVIANT PEER RELATIONS (INDIRECT TARGETS). In the parallel process model for Aim 2, the *a-path* is identical to that for Aim 1. The "outcome" model is nearly identical, the only difference being that the "outcomes" are indirect targets of treatment, behavioral regulation and peer relations. The b-path coefficient represents the association between the during-treatment slope for parent management and the 9- and 12-months post-treatment levels of behavioral regulation and peer relations.

AIM 3: DETERMINE WHETHER BEHAVIORAL REGULATION & DEVIANT PEER RELATIONS (INDIRECT TARGETS) MEDIATE THE EFFECT OF PARENT MANAGEMENT SKILLS (DIRECT TARGET) ON YOUTH SUBSTANCE USE & BEHAVIOR PROBLEMS (ULTIMATE OUTCOMES). Aim 3 uses the same approach, with one key difference: rather than treatment condition, the initial variable is parent management (the direct target of treatment) and, as such, there are repeated measurements. The *a-path* represents the effect of parent management on behavioral regulation and deviant peer relations. With both measured longitudinally, this takes the form of the during-treatment slope for parent management predicting the during-treatment slope for behavioral regulation and deviant peer relations. Although this could confound timing and sequencing of a-path effects, the results of Aim 2 will have established the extent to which there is evidence supporting a causal association between the direct and indirect targets of treatment. The outcome model is identical to that for Aim 1. The *b-path*, holding constant the effect of parent management, is the effect of the during-treatment slopes for behavioral regulation and peer relations on the post-treatment levels of substance use and behavior problems.

**STATISTICAL POWER FOR MEDIATED EFFECTS.** The proposed mediation models include estimates of: (1) the effect of the initial variable on the hypothesized mediator (α-path), (2) the effect of the hypothesized mediator on the outcome (β-path), and (3) the mediated effect (αβ). Using Monte Carlo simulations implemented in Mplus,  $^{214-215}$  power is determined by the percentage of replications with a significant effect for the path of interest. Using covariance algebra provided by Thoemmes et al.,  $^{215}$  parameters (path coefficients, variances, residuals) were tailored to reflect α- and β-paths with small-to-medium ( $R^2 = .07$ ) effects. For each model, sample size, conservatively assuming 10% attrition, was 155, with 10000 replications from the population. For a-path, power was >.90 to detect a small-to-medium effect of the initial variable on the mediator. For β-path, power was .85 to detect a small-to-medium effect of intermediate targets on ultimate outcomes. For the mediated effect, power was .83. This estimate is conservative due to the simulation's Sobell *SE* method. As an upper bound on power, and based on simulations using the proposed asymmetric *SE* method, Fritz and MacKinnon<sup>216</sup> found a sample of *N*=74 sufficient for .80 power to detect medium effects for α- and β-paths.

# **ATTRITION AND MISSING DATA**

Participants will be retained in research measurement independent of CM/CM+ participation following intent-to-treat principles.<sup>217</sup> Along with this, the successful participant tracking and retention protocols used in OSLC research will minimize missing data. However, because some data will inevitably be missing, methods recommended by Schafer and Graham<sup>218</sup> will evaluate assumptions and guide analyses. Three steps will be used: (1) For a small proportion of missing data with evidence of Missing at Random (MAR), data will be analyzed using the estimation procedures described above. (2) For a non-trivial amount of missing data and evidence of MAR, multiple imputation for repeated measurements will generate complete data.<sup>219</sup> (3) For a non-random missing data mechanism, pattern mixture models will identify and control its effects.<sup>203–204</sup>

# **BIBLIOGRAPHY & REFERENCES CITED**

- 1. Chamberlain, P., & Reid J. (1987). Parent observation and report of child symptoms. *Behavioral Assessment*, 9, 97-109.
- 2. Forgatch, M. S., & Patterson, G. R. (2010). *Parent Management Training-Oregon Model: An intervention for antisocial behavior in children and adolescents.* In J. R. Weisz & A. E. Kazdin (Eds.), Evidence-based psychotherapies for children and adolescents (2<sup>nd</sup> ed., pp. 159-178). New York: Guilford.
- 3. Strada, M. J., Donohue, B., & Lefforge, N. L. (2006). Examination of ethnicity in controlled treatment outcome studies involving adolescent substance abusers: A comprehensive literature review. *Psychology of Addictive Behaviors, 20*, 11–27.
- 4. Tienda, M., & Mitchell, F. (2006). *National Research Council Panel on Hispanics in the United States*. Washington, DC: National Academies Press.
- 5. Santisteban, D. A., Coatsworth, J. D., Perez-Vidal, A., Kurtines, W. M., Schwartz, S. J., LaPierre, A., et al. (2003). Efficacy of brief strategic family therapy in modifying Hispanic adolescent behavior problems and substance use. *Journal of Family Psychology, 17*, 121–133.
- 6. Szapocznik, J., Perez-Vidal, A., Brickman, A. L., Foote, F. H., Santisteban, D., Hervis, O., & Kurtines, W. M. (1988). Engaging adolescent drug abusers and their families in treatment: A strategic structural systems approach. *Journal of Consulting and Clinical Psychology*, *56*, 552–557.
- 7. Waldron, H. B., Slesnick, N., Brody, J. L., Turner, C. W., & Peterson, T. R. (2001). Treatment outcomes for adolescent substance abuse at 4- and 7-month assessments. *Journal of Consulting and Clinical Psychology*, 69, 802–813.
- 8. Waldron, H. B., & Turner, C. W. (2008). Evidence-based psychosocial treatments for adolescent substance abuse. *Journal of Clinical Child and Adolescent Psychology*, *37*, 238-261.
- 9. Robbins, M. S., Szapocznik, J., Dillon, F. R., Turner, C. W., Mitrani, V. B., & Feaster D. J. (2008). The efficacy of structural ecosystems therapy with drug-abusing/dependent African American and Hispanic American adolescents. *Journal of Family Psychology*, 22, 51-61.
- 10. Huey, S., & Polo, A. (2008). Evidence-based psychosocial treatments for ethnic minority youth: A review and meta-analysis. *Journal of Clinical Child and Adolescent Psychology*, 37, 262-301.
- 11. McLellan A. T., Carise D., & Kleber H. D. (2003). Can the national addiction treatment infrastructure support the public's demand for quality care? *Journal of Substance Abuse Treatment*, 25, 117-121.
- 12. Substance Abuse and Mental Health Services Administration. (2014). *National survey of substance abuse treatment services (N-SSATS): 2013. Data on substance abuse treatment facilities.* Rockville, MD: U.S. Department of Health and Human Services.
- Hogue, A., Henderson, C. E., Ozechowski, T. J., & Robbins, M. S. (2014). Evidence base on outpatient behavioral treatments for adolescent substance use: Updates and recommendations 2007–2013. *Journal of Clinical Child and Adolescent Psychology*, 43(5):695-720.
- 14. Grella, C. E., Joshi, V., & Hser, Y. I. (2004). Effects of comorbidity on treatment processes and outcomes among adolescents in drug treatment programs. *Journal of Child and Adolescent Substance Abuse*, *13*, 13-31.
- 15. Williams, R. J., & Chang, S. Y. (2000). A comprehensive and comparative review of adolescent substance abuse treatment outcome. *Clinical Psychology: Science and Practice*, 7, 138-166.
- 16. Winters, K. C., Botzet, A. M., & Fahnhorst, T. (2011). Advances in adolescent substance abuse treatment. *Current Psychiatry Reports*, *13*, 416-421.
- 17. MacKinnon, D. P., & Fairchild, A. J. (2009). Current directions in mediation analysis. *Current Directions in Psychological Science*, 18, 16-20.
- 18. Pirlott, A. G., & MacKinnon, D. P. (2016). Design approaches to experimental mediation. Journal of Experimental Social Psychology, 66, 29-38.
- 19. Waldron, H. B., & Turner, C. W. (2008). Evidence-based psychosocial treatments for adolescent substance abuse. *Journal of Clinical Child and Adolescent Psychology*, 37, 238-261.

- 20. McCart, M. R., & Sheidow, A. J. (2016). Evidence-based psychosocial treatments for adolescents with disruptive behavior. *Journal of Clinical Child and Adolescent Psychology*, 45(5), 529-563.
- 21. Brown, S. A., & Abrantes, A. M. (2006). Substance use disorders. In. D. A. Wolfe & E. J. Mash (Eds.). *Behavioral and emotional disorders in adolescents*. Guildford: New Nork, NY.
- 22. Cleveland, M. J., Feinberg, M. E., Bontempo, D. E., & Greenberg, M. T. (2008). The role of risk and protective factors in substance use across adolescence. *Journal of Adolescent Health*, 43, 157-164.
- 23. Bryck, R. L., & Fisher, P. A. (2012). Training the brain: Practical applications of neural plasticity from the intersection of cognitive neuroscience, developmental psychology, and prevention science. *American Psychologist*, 67(2), 87–100.
- 24. Diamond, A., & Lee, K. (2011). Interventions shown to aid executive function development in children 4 to 12 years old. *Science*, 333, 959–964.
- 25. McCart, M. R., Priester, P., Davies, W. H., & Azen, R. (2006). Differential effectiveness of behavioral parent-training and cognitive-behavioral therapy for antisocial youth: A meta-analysis. *Journal of Abnormal Child Psychology*, 34, 527-543.
- 26. Burrus, B., Leeks, K. D., Sipe, T. A., Dolina, S., Soler, R., Elder, R., ...Achrekar, A. (2012). Person-to-person interventions targeted to parents and other caregivers to improve adolescent health: A community guide systematic review. *American Journal of Preventive Medicine*, *42*(3), 316-326.
- 27. Chang, H., Shaw, D. S., Dishion, T. J., Gardner, F., & Wilson, M. N. (2015). Proactive parenting and children's effortful control: Mediating role of language and indirect intervention effects. *Social Development*, *24*(1), 206–223.
- 28. Jankowski, K. F., Bruce, J., Beauchamp, K. G., Roos, L. E., Moore, W. E., & Fisher, P. A. (2016). Preliminary evidence of the impact of early childhood maltreatment and a preventive intervention on neural patterns of response inhibition in early adolescence. *Developmental Science*.
- 29. McDermott, J. M., Westerlund, A., Zeanah, C. H., Nelson, C. A., & Fox, N. A. (2012). Early adversity and neural correlates of executive function: Implications for academic adjustment. *Developmental Cognitive Neuroscience*, 2(Supplement 1), S59–S66.
- 30. Castellanos-Ryan, N., Séguin, J. R., Vitaro, F., Parent, S., & Tremblay, R. E. (2013). Impact of a 2-year multimodal intervention for disruptive 6-year-olds on substance use in adolescence: Randomised controlled trial. *British Journal of Psychiatry*, 203(3), 188–195.
- 31. DeLay, D., Ha, T., Van Ryzin, M. J., Winter, C., & Dishion, T. J. (2016). Changing friend selection in middle school: A social network analysis of a randomized intervention study designed to prevent adolescent problem behavior. *Prevention Science*, 17(3), 285-294.
- 32. Azrin, N. H., Acierno, R., Kogan, E. S., Donohue, B., Besalel V. A., & McMahon, P. T. (1996). Follow-up results of supportive versus behavioral therapy for illicit drug use. *Behaviour Research and Therapy*, 34, 41-46.
- 33. Donohue, B., & Azrin, N. H. (2001). Family behavior therapy. In E. F. Wagner, H. B. Waldron (Eds.), *Innovations in adolescent substance abuse interventions*. New York, NY: Pergamon Press.
- 34. Henggeler, S. W., McCart, M. R., Cunningham, P. B., & Chapman, J. E. (2012). Enhancing the effectiveness of juvenile drug courts by integrating evidence-based practices. *Journal of Consulting and Clinical Psychology*, 80(2), 264-275. PMCID: PMC22309470.
- 35. Henggeler, S. W., Chapman, J. E., Rowland, M. D., et al. (2007). If you build it, they will come: Statewide practitioner interest in CM for youths. *Journal of Substance Abuse Treatment*, 32, 121-131. PMID: 17306721.
- 36. Henggeler, S. W., Chapman, J. E., Rowland, M. D., et al. (2008). Statewide adoption and initial implementation of contingency management for substance abusing adolescents. *Journal of Consulting and Clinical Psychology*, *76*, 556-567. PMCID: PMC2603081.
- 37. McCart, M. R., Henggeler, S. W., Chapman, J. E., & Cunningham, P. B. (2012). System-level effects of integrating a promising treatment into juvenile drug courts. *Journal of Substance Abuse Treatment*, 43, 231-243. PMCID: PMC3309115.
- 38. Godley, S. H., Garner, B. R., Passetti, L. L., Funk, R. R., Dennis, M. L., & Godley, M. D. (2010). Adolescent outpatient treatment and continuing care: Main findings from a randomized clinical trial. *Drug and Alcohol Dependence*, *110*, 44-54.
- 39. Substance Abuse and Mental Health Services Administration. (2014). Results from the 2013 National Survey on Drug Use and Health. Rockville, MD: U.S. Department of Health and Human Services.

- 40. Alford, G. S., Koehler, R. A., & Leonard, J. (1991). Alcoholics Anonymous-Narcotics Anonymous model inpatient treatment of chemically dependent adolescents: A 2-year outcome study. *Journal of Studies on Alcohol*, *52*(2), 118-126.
- 41. Chan, Y. F., Dennis, M. L., & Funk, R. R. (2008). Prevalence and comorbidity of major internalizing and externalizing problems among adolescents and adults presenting to substance abuse treatment. *Journal of Substance Abuse Treatment*, 34(1), 14-24.
- 42. Crowley, T. J., Mikulich, S. K., MacDonald, M., Young, S. E., & Zerbe, G. O. (1998). Substance-dependent, conduct-disordered adolescent males: Severity of diagnosis predicts 2-year outcome. *Drug and Alcohol Dependence*, 49(3), 225-237.
- 43. Henggeler, S. W., Clingempeel, W. G., Brondino, M. J., & Pickrel, S. G. (2002). Four-year follow-up of MST with substance-abusing and dependent juvenile offenders. *Journal of the American Academy of Child and Adolescent Psychiatry*, 41(7), 868-874.
- 44. Myers, M. G., Stewart, D. G., & Brown, S. A. (1998). Progression from conduct disorder to antisocial personality disorder following treatment for adolescent substance abuse. *American Journal of Psychiatry*, 155(4), 479-485.
- 45. Ringel, J. S., Ellickson, P. L., & Collins, R. L. (2007). High school drug use predicts job-related outcomes at age 29. *Addictive Behaviors*, 32(3), 576-589.
- 46. National Institute on Drug Abuse. *Trends and Statistics*. (2015), Retrieved from http://www.drugabuse.gov/related-topics/trends-statistics.
- 47. Diamond, G., & Josephson, A. (2005). Family-based treatment research: a 10-year update. Journal of the American Academy of Child and Adolescent Psychiatry, 44(9), 872-887.
- 48. Tanner-Smith, E. E., Wilson, S. J., & Lipsey, M. W. (2013). The comparative effectiveness of outpatient treatment for adolescent substance abuse: A meta-analysis. *Journal of Substance Abuse Treatment*, 44, 145-158.
- 49. Robbins, M. S., Feaster, D. J., Horigian, V. E., et al. (2011). Brief strategic family therapy versus treatment as usual: Results of a multisite randomized trial for substance using adolescents. *Journal of Consulting and Clinical Psychology*, 79(6), 713-727.
- 50. Santisteban, D. A., Coatsworth, J. D., Perez-Vidal, A., et al. (2003). Efficacy of brief strategic family therapy in modifying Hispanic adolescent behavior problems and substance use. *Journal of Family Psychology*, 17, 121-133.
- Journal of Family Psychology, 17, 121-133.
  51. Slesnick, N., & Prestopnik, J. L. (2009). Comparison of family therapy outcome with alcoholabusing, runaway adolescents. Journal of Marital and Family Therapy, 35(3), 255-277.
- 52. Waldron, H. B., Ślesnick, N., Brody, J. L., Turner, C. W., & Peterson, T. R. (2001). Treatment outcomes for adolescent substance abuse at 4- and 7-month assessments. *Journal of Consulting and Clinical Psychology*, 69, 802-813.
- 53. Liddle, H. A., Dakof, G. A., Diamond, G., Parker, K., Barrett, K., & Tejeda, M. (2001). Multidimensional family therapy for adolescent drug abuse: Results of a randomized clinical trial. *American Journal of Drug and Alcohol Abuse*, 27, 652-687.
- 54. Liddle, H. A., Rowe, C. L., Ďakof, G. A., Henderson, C. E., & Greenbaum, P. E. (2009). Multidimensional family therapy for young adolescent substance abuse: Twelve-month outcomes of a randomized controlled trial. *Journal of Consulting and Clinical Psychology*, 77(1), 12-25.
- 55. Henggeler, S. W., Halliday-Boykins, C., Cunningham, P. B., Randall, J., Shapiro, S. B., & Chapman, J. E. (2006). Juvenile drug court: Enhancing outcomes by integrating evidence-based treatments. *Journal of Consulting and Clinical Psychology*, *74*, 42-54.
- 56. Kaminer, Y., Burleson, J. A., & Goldberger, R. (2002). Cognitive-behavioral coping skills and psychoeducation therapies for adolescent substance abuse. *Journal of Nervous and Mental Disease*, 190, 737-745.
- 57. Hunter, S. B., Ramchand, R., Griffin, B. A., Suttorp, M. J., McCaffrey, D., & Morral, A. (2012). The effectiveness of community-based delivery of an evidence-based treatment for adolescent substance use. *Journal of Substance Abuse Treatment*, *43*(2), 211-220.
- 58. Martin, G., & Copeland, J. (2008). The adolescent cannabis check-up: Randomized trial of a brief intervention for young cannabis users. *Journal of Substance Abuse Treatment*, 34, 407–414.
- 59. Walker, D. D., Stephens, R., Roffman, R., DeMarce, J., Lozano, B., Towe, S., & Berg, B. (2011). A randomized controlled trial of motivational enhancement therapy with nontreatment-seeking adolescent cannabis users: A further test of the Teen Marijuana Check-Up. *Psychology of Addictive Behaviors*, 25, 474–484.

- 60. Dube, S. R., Felitti, V. J., Dong, M., Chapman, D. P, Giles, W. H., & Anda R. F. (2003). Childhood abuse, neglect, and household dysfunction and the risk of illicit drug use: the adverse childhood experiences study. *Pediatrics*, *111*(3), 564-572.
- 61. Skeer, M., McCormick, M. C., Normand, S. L., Buká, S. L., & Gilman, S. E. (2009). A prospective study of familial conflict, psychological stress, and the development of substance use disorders in adolescence. *Drug and Alcohol Dependence*, 104(1-2), 65-72.
- 62. Dowell, K. A., & Ogles, B. M. (2010). The effects of parent participation on child psychotherapy outcome: A meta-analytic review. *Journal of Clinical Child and Adolescent Psychology*, 39, 151-162.
- 63. Bender, K., Tripodi, S. J., Sarteschi, C., & Vaughn, M. G. (2011). A meta-analysis of interventions to reduce adolescent cannabis use. *Research on Social Work Practice*, *21*,153-164.
- 64. Bullock, J. G., Green, D. P., & Ha, S. E. (2010). Yes, but what's the mechanism? (Don't expect an easy answer). *Journal of Personality and Social Psychology*, 98, 550–558.
- 65. Howell, J. C. (2008). Preventing and reducing juvenile delinquency: A comprehensive framework. Thousand Oaks, CA: Sage.
- 66. Liberman, A. M. (2008). The long view of crime: A synthesis of longitudinal research. New York, NY: Springer.
- 67. Loeber, R., Burke, J. & Pardini, D. A. (2009). Perspectives on oppositional defiant disorder, conduct disorder, and psychopathic features. *Journal of Child Psychology and Psychiatry*.
- 68. Casey, B. J., & Jones, R. M. (2010). Neurobiology of the adolescent brain and behavior: Implications for substance use disorders. *Journal of the American Academy of Child and Adolescent Psychiatry*, 49, 1189–1201.
- 69. Chambers, R. A., Taylor, J. R., & Potenza, M. N. (2003). Developmental neurocircuitry of motivation in adolescence: A critical period of addiction vulnerability. *American Journal of Psychiatry*, 160, 1041–52.
- 70. Ernst, M., Pine, D. S., & Hardin, M. (2006). Triadic model of the neurobiology of motivated behavior in adolescence. *Psychological Medicine: A Journal of Research in Psychiatry and the Allied Sciences*, 36, 299–312.
- 71. Steinberg, L. (2008). A social neuroscience perspective on adolescent risk-taking. *Developmental Review*, 28, 78–106.
- 72. Byrnes, J. P., Miller, D. C., & Schafer, W. D. (1999). Gender differences in risk taking: A meta-analysis. *Psychological Bulletin*, *125*, 367–83.
- 73. Leigh, B. C. (1999). Peril, chance, adventure: Concepts of risk, alcohol use, and risky behavior in young adults. *Addiction*, *94*, 371–83.
- Lejuez, C. W., Read, J. P., Kahler, C. W., et al. (2002). Evaluation of a behavioral measure of risk-taking: The Balloon Analogue Risk Task (BART). Journal of Experimental Psychology: Applied, 8, 75–84.
- 75. Casey, B. J., Tottenham, N., & Fossella, J. (2002). Clinical, imaging, lesion, and genetic approaches toward a model of cognitive control. *Developmental Psychobiology*, 40, 237–54.
- 76. Durston, S., Thomas, K. M., Yang, Y., Ulug, A. M., Zimmerman, R. D., & Casey, B. J. (2002). A neural basis for the development of inhibitory control. *Developmental Science*, *5*, F9–F16.
- 77. Aklin, W. M., Lejuez, C. W., Zvolensky, M. J., Kahler, C. W., & Gwadz, M. (2005). Evaluation of behavioral measures of risk taking propensity with inner city adolescents. *Behaviour Research and Therapy*, 43, 215–28.
- 78. Deckel, A. W., & Hesselbrock, V. (1996). Behavioral and cognitive measurements predict scores on the MAST: A 3-year prospective study. *Alcoholism: Clinical and Experimental Research*, 20, 1173–1178.
- 79. Dubow, E. F., Boxer, P., & Huesmann, L. R. (2008). Childhood and adolescent predictors of early and middle adulthood alcohol use and problem drinking: The Columbia County Longitudinal Study. *Addiction*, 103, 36–47.
- 80. Johnson, C. A., Xiao, L., Palmer, P., et al. (2008). Affective decision-making deficits, linked to a dysfunctional ventromedial prefrontal cortex, revealed in 10th grade Chinese adolescent binge drinkers. *Neuropsychologia*, 46,714–26.
- 81. Lejuez, C. W., Aklin, W., Daughters, S., Zvolensky, M., Kahler, C., & Gwadz, M. (2007). Reliability and validity of the youth version of the Balloon Analogue Risk Task (BART–Y) in the assessment of risk-taking behavior among inner-city adolescents. *Journal of Clinical Child and Adolescent Psychology*, 36, 106–11.

- 82. MacPherson, L., Magidson, J. F., Reynolds, E. K., Kahler, C. W., & Lejuez, C. W. (2010). Changes in sensation seeking and risk-taking propensity predict increases in alcohol use among early adolescents. *Alcoholism: Clinical and Experimental Research*, 34, 1400–1408.
- 83. Pears, K. C., Capaldi, D. M., & Owen, L. D. (2007). Substance use risk across three generations: The roles of parent discipline practices and inhibitory control. *Psychology of Addictive Behaviors*, *21*, 373–86.
- 84. Wills, T. A., & Stoolmiller, M. (2002). The role of self-control in early escalation of substance use: A time-varying analysis. *Journal of Consulting and Clinical Psychology*, 70, 986–97.
- 85. Williams, L. R., Fox, N. A., Lejuez, C. W., et al. (2010). Early temperament, propensity for risk-taking and adolescent substance-related problems: A prospective multi-method investigation. *Addictive Behaviors*, *35*, 1148–51.
- 86. Bowden-Jones, H., McPhillips, M., Rogers, R., Hutton, S., & Joyce, E. (2005). Risk-taking on tests sensitive to ventromedial prefrontal cortex dysfunction predicts early relapse in alcohol dependency: A pilot study. *Journal of Neuropsychiatry and Clinical Neurosciences*, *17*, 417–420.
- 87. Krishnan-Sarin, S., Reynolds, B., Duhig, A. M., et al. (2007). Behavioral impulsivity predicts treatment outcome in a smoking cessation program for adolescent smokers. *Drug and Alcohol Dependence*, 88, 79–82.
- 88. Passetti, F., Clark, L., Mehta, M. A., Joyce, E., & King, M. (2008). Neuropsychological predictors of clinical outcome in opiate addiction. *Drug and Alcohol Dependence*, *94*, 82–91.
- 89. Schmitz, J. M., Mooney, M. E., Green, C. E., et al. (2009). Baseline neurocognitive profiles differentiate abstainers and non-abstainers in a cocaine clinical trial. *Journal of Addictive Diseases*, 28, 250–7.
- 90. Dodge, K. A., Dishion, T. J., & Lansford, J. E. (Eds.). (2007). Deviant peer influences in programs for youth: Problems and solutions. New York, NY: Guilford Press.
- 91. Andrews, J. A., Tildesley, E., Hops, H., & Li, F. (2002). The influence of peers on young adult substance use. *Health Psychology*, *21*(4), 349-357.
- 92. Fleming, C. B., Catalano, R. F., Haggerty, K. P., & Abbott, R. D. (2010). Relationships between level and change in family, school, and peer factors during two periods of adolescence and problem behavior at age 19. *Journal of Youth and Adolescence*, 39(6), 670-682.
- 93. Patterson, G. R., Dishion, T. J., & Yoerger, K. (2000). Adolescent growth in new forms of problem behavior: Macro- and micro-peer dynamics. *Prevention Science*, 1(1), 3-13.
- 94. Huey, S., J., Henggeler, S. W., Brondino, M. J., & Pickrel, S. G. (2000). Mechanisms of change in Multisystemic Therapy: Reducing delinquent behavior through therapist adherence, and improved family and peer functioning. *Journal of Consulting and Clinical Psychology*, 68(3), 451-467.
- 95. Eddy, J. M., & Chamberlain, P. (2000). Family management and deviant peer association as mediators of the impact of treatment condition on youth antisocial behavior. *Journal of Consulting and Clinical Psychology*, 68(5), 857-863.
- 96. Van Ryzin, M. J., & Leve, L. D. (2012). Affiliation with delinquent peers as a mediator of the effects of Multidimensional Treatment Foster Care for delinquent girls. *Journal of Consulting and Clinical Psychology*, 80(4), 588-596.
- 97. Dishion, T. J., Bullock, B. M., & Granic, I. (2002). Pragmatism in modeling peer influence: Dynamics, outcomes, and change processes. *Development and Psychopathology*, *14*(4), 969-981.
- 98. Hoge, R. D., Guerra, N. G., & Boxer, P. (Eds.). (2008). Treating the juvenile offender. New York, NY: Guilford Press.
- 99. Patterson, G. R. (2002). The early developmental of coercive family process. In J. B. Reid, G. R. Patterson & J. Snyder (Eds.), *Antisocial behavior in children and adolescents: A developmental analysis and model for intervention* (pp. 25-44). Washington DC: American Psychological Association.
- 100. Crossley, I. A., & Buckner, J. C. (2012). Maternal-related predictors of self-regulation among low-income youth. *Journal of Child and Family Studies*, *21*, 217–27.
- 101. Finkenauer, C., Engels, R. C. M. E., & Baumeister, R. F. (2005). Parenting behaviour and adolescent behavioural and emotional problems: The role of self-control. *International Journal of Behavioral Development*, 29, 58–69.
- 102. Moilanen, K. L., Shaw, D. S., & Fitzpatrick, A. (2010). Self-regulation in early adolescence: Relations with mother-son relationship quality and maternal regulatory support and antagonism. *Journal of Youth and Adolescence*, 39, 1357–67.

- 103. Simons, L. G., Sutton, T. E., Simons, R. L., Gibbons, F. X., & Murry, V. M. (2016). Mechanisms that link parenting practices to adolescents' risky sexual behavior: A test of six competing theories. *Journal of Youth and Adolescence*, 45, 255–70.
- 104. Fosco, G. M., Frank. J. L., Stormshak, E. A., & Dishion, T. J. (2013). Opening the "Black Box": Family check-up intervention effects on self-regulation that prevents growth in problem behavior and substance use. *Journal of School Psychology*, *51*, 455–68.
- 105. Koning, I. M., Maric, M., MacKinnon, D., Vollebergh, W. A. M. (2015). Effects of a combined parent–student alcohol prevention program on intermediate factors and adolescents' drinking behavior: A sequential mediation model. *Journal of Consulting and Clinical Psychology*, 83, 719–27.
- 106. Mason, W. A., Fleming, C. B., Ringle, J. L., Thompson, R. W., Haggerty, K. P., & Snyder, J. J. (2015). Reducing risks for problem behaviors during the high school transition: Proximal outcomes in the Common Sense Parenting trial. *Journal of Child and Family Studies*, 24, 2568–78.
- 107. Letourneau, E. J., McCart, M. R., Sheidow, A. J., & Mauro, P. M. (2017). First evaluation of a contingency management intervention addressing adolescent substance use and sexual risk behaviors: Risk reduction therapy for adolescents. *Journal of Substance Abuse Treatment*, 72, 56-65.
- 108. Godley, M. D., Godley, S. H., Dennis, M. L., Funk, R. R., Passetti, L. L., & Petry, N. M. (2014). A randomized trial of assertive continuing care and contingency management for adolescents with substance use disorders. *Journal of Consulting and Clinical Psychology*, 82, 40-51.
- 109. Prendergast, M., Podus, D., Finney, J., Greenwell, L., & Roll, J. (2006). Contingency management for treatment of substance use disorders: A meta-analysis. *Addiction*, 101, 1546-1560.
- 110. Benishek, L. A., Dugosh, K. L., Kirby, K. C., Matejkowski, J., Clements, N. T., Seymour, B. L., & Festinger, D. S. (2014). Prize-based contingency management for the treatment of substance abusers: A meta-analysis. *Addiction*, 109, 1426-1436.
- 111. Loeber, R., Farrington, D. P., Stouthamer-Loeber, M., & Van Kammen, W. B. (1998). *Antisocial behavior and mental health problems: Explanatory factors in childhood and adolescence*. Mahwah, NJ: Lawrence Erlbaum Associates.
- 112. Kazdin, A. E., & Nock, M. K. (2003). Delineating mechanisms of change in child and adolescent therapy: Methodological issues and research recommendations. *Journal of Child Psychology and Psychiatry*, *44*, 1116-1129.
- 113. Higa-McMillan, C. K., Francis, S. E., Rith-Najarian, L., & Chorpita, B. F. (2016). Evidence base update: 50 years of research on treatment for child and adolescent anxiety. *Journal of Clinical Child and Adolescent Psychology*, *45*, 91-113.
- 114. Fristad, M. A., & MacPherson, H. A. (2014). Evidence-based psychosocial treatments for child and adolescent bipolar spectrum disorders. *Journal of Clinical Child and Adolescent Psychology*, 43, 339-355.
- 115. Glenn, C. R., Franklin, J. C., & Nock, M. K. (2015). Evidence-based psychosocial treatments for self-injurious thoughts and behaviors in youth. *Journal of Clinical Child and Adolescent Psychology*, 44, 1-29.
- 116. Stanger, C., Budney, A. J., & Bickel, W. K. (2013). A developmental perspective on neuroeconomic mechanisms of contingency management. *Psychology of Addictive Behaviors*, 27, 403–15.
- 117. Henggeler, S. W., Sheidow, A. J., Cunningham, P. B., Donohue, B., & Ford, J. D. (2008). Promoting the implementation of an evidence-based intervention for adolescent marijuana abuse in community settings: Testing the use of intensive quality assurance. *Journal of Clinical Child and Adolescent Psychology*, 37, 682-689.
- 118. Henggeler, S. W. (2011). Efficacy studies to large-scale transport: The development and validation of multisystemic therapy programs. *Annual Review of Clinical Psychology*, 7, 351-381.
- 119. Bruce, J., Fisher, P. A., Graham, A. M., Moore, W. E., Peake, S. J., & Mannering, A. M. (2013). Patterns of brain activation in foster children and nonmaltreated children during an inhibitory control task. *Development and Psychopathology*, *25*, 931–941.
- 120. Bruce, J., Tarullo, A. R., & Gunnar, M. R. (2009). Disinhibited social behavior among internationally adopted children. *Development and Psychopathology*, *21*, 157–171.
- 121. Davis, E. P., Bruce, J., Snyder, K., & Nelson, C. A. (2003). The X-trials: Neural correlates of an inhibitory control task in children and adults. *Journal of Cognitive Neuroscience*, *15*(3), 432–443.

- 122. Pears, K. C., Fisher, P. A., Bruce, J., Kim, H. K., Yoerger, K. (2010). Early elementary school adjustment of maltreated children in foster care: The roles of inhibitory control and caregiver involvement. *Child Development*, *81*(5), 1550–1564.
- 123. Roos, L. E., Pears, K. C., Bruce, J., Kim, H. K., & Fisher, P. A. (2015). Impulsivity and the association between the feedback-related negativity and performance on an inhibitory control task in young at-risk children. *Psychophysiology*, *52*, 704–713.
- 124. Bruce, J., McDermott, J. M., Fisher, P. A., & Fox, N. A. (2009). Using behavioral and electrophysiological measures to assess the effects of a preventive intervention: A preliminary study with preschool-aged foster children. *Prevention Science*, 10, 129–140.
- 125. Graham, A. M., Yockelson, M., Kim, H. K., Bruce, J., Pears, K. C., & Fisher P. A. (2012). Effects of maltreatment and early intervention on diurnal cortisol slope across the start of school: A pilot study. *Child Abuse and Neglect*, *36*, 660–670.
- 126. McDermott, J. M., Pears, K. C., Bruce, J., et al. (2015). Improving kindergarten readiness in children with developmental disabilities: Changes in neural correlates of response monitoring. Manuscript revised and resubmitted for publication.
- 127. Henggeler, S. W., Letourneau, E. J., Chapman, J. E., Borduin, C. M., Schewe, P. A., & McCart, M. R. (2009). Mediators of change for multisystemic therapy with juvenile sexual offenders. *Journal of Consulting and Clinical Psychology*, 77(3), 451-462. PMCID: PMC2744326.
- 128. Leve, L. D., & Chamberlain, P. (2007). A randomized evaluation of Multidimensional Treatment Foster Care: Effects on school attendance and homework completion in juvenile justice girls. *Research on Social Work Practice*, 17(6), 657-663.
- 129. Azrin, N. H., Donohue, B., Besalel, V. A., Kogan, E. S., & Acierno, R. (1994). Youth drug abuse treatment: A controlled outcome study. *Journal of Child and Adolescent Substance Abuse*, *3*, 1-16.
- 130. Azrin, N. H., McMahon, P. T., Donohue, B., et al. (1994). Behavior therapy for drug abuse: A controlled treatment outcome study. *Behaviour Research and* Therapy, 32(8), 857-866.
- 131. McCart, M. R., Sheidow, A. J., & Letourneau, E. J. (2014). Risk Reduction Therapy for Adolescents (RRTA): Targeting substance use and HIV/STI-risk behaviors. *Cognitive and Behavioral Practice*, *21*, 161-175. PMCID: PMC4235161.
- 132. Merrill, M. D. (2002). First principles of instruction. *Educational Technology Research and Development*, 50, 43-59.
- 133. Reigeluth, C. M. (1999). Instructional-design theories and models: A new paradigm of instructional theory. Vol II. Lawrence Erlbaum: Mahwah, NJ.
- 134. Burke, L. A., & Hutchins, H. M. (2007). Training transfer: An integrative literature review. *Human Resource Development Review*, *6*, 263-296.
- 135. Petry, N. M. (2010). Contingency management treatments: Controversies and challenges. *Addiction*, 105, 1507-1509.
- 136. Roll, J. M., & Shoptaw, S. (2006). Contingency management for the treatment of methamphetamine abuse: Schedule effects. *Psychiatry Research*, *144*, 91-93.
- 137. Henggeler, S. W., Melton, G. B., Brondino, M. J., Scherer, D. G., & Hanley, J. H. (1997). Multisystemic therapy with violent and chronic juvenile offenders and their families: The role of treatment fidelity in successful dissemination. *Journal of Consulting and Clinical Psychology*, 65(5), 821-833.
- 138. Borduin, C. M., Mann, B. J, Cone, L. T., et al. (1995). Multisystemic treatment of serious juvenile offenders: Long-term prevention of criminality and violence. *Journal of Consulting and Clinical Psychology*, 63(4), 569-578.
- 139. Henggeler, S. W., Melton, G. B., & Smith, L. A. (1992). Family preservation using Multisystemic therapy: An effective alternative to incarcerating serious juvenile offenders. *Journal of Consulting and Clinical Psychology*, 60, 953-961.
- 140. Rowland, M. D., Halliday-Boykins, C., Henggeler, S. W., et al. (2005). A randomized trial of Multisystemic therapy with Hawaii's Felix class youths. *Journal of Emotional and Behavioral Disorders*, 3, 13-23.
- 141. Chamberlain, P., & Reid J. (1998). Comparison of two community alternatives to incarceration for chronic juvenile offenders. *Journal of Consulting and Clinical Psychology*, *6*(4), 624-633.
- 142. Leve, L. D., Chamberlain, P., & Reid, J. B. (2005). Intervention outcomes for girls referred from juvenile justice: Effects on delinquency. *Journal of Consulting and Clinical Psychology*, 73, 1181-1185.
- 143. Holth, P., Torsheim, T., Sheidow, A. J., Ogden, T., & Henggeler, S. W. (2011). Intensive quality assurance of therapist adherence to contingency management for adolescent substance use problems. *Journal of Child and Adolescent Substance Abuse*, 20, 289-313.

- 144. Henggeler, S. W., Chapman, J. E., Rowland, M. D., Sheidow, A. J., & Cunningham, P. B. (2013). Evaluating training methods for transporting contingency management to therapists. *Journal of Substance Abuse Treatment*, *45*, 466-474. PMCID: PMC3805110.
- 145. Petry, N. M., Alessi, S. M., & Ledgerwood, D. M. (2012). Contingency management delivered by community therapists in outpatient settings. *Drug and Alcohol Dependence*, *122*, 86-92.
- 146. Petry, N. M., Alessi, S. M., & Ledgerwood, D. M. (2012). A randomized trial of contingency management delivered by community therapists. *Journal of Consulting and Clinical Psychology*, 80(2), 286-298.
- 147. Rash, C. J., Dephilippis, D., McKay, J. R., Drapkin, M., & Petry, N. M. (2013). Training workshops positively impact beliefs about contingency management in a nationwide dissemination effort. *Journal of Substance Abuse Treatment*, 45(3), 306-312.
- 148. Schoenwald, S. K., Carter, R. E., Chapman, J. E., & Sheidow, A. J. (2008). Therapist adherence and organizational effects on change in youth behavior problems one year after multisystemic therapy. *Administration and Policy in Mental Health and Mental Health Services Research*, 35(5), 379-394.
- 149. Martinez, C., & Eddy, M. (2005). Effects of culturally adapted Parent Management Training on Latino youth behavioral health outcomes. *Journal of Consulting and Clinical Psychology*, 73(4), 1-851.
- 150. Martinez, C. R., McClure, H. H., & Eddy, J. E. (2009). Language brokering contexts and behavioral and emotional adjustment among Latino parents and adolescents. *Journal of Early Adolescence*, 5, 71-98.
- 151. Dennis, M. L., Titus, J. C., White, M., Unsicker, J., & Hodgkins, D. (2002). *Global Appraisal of Individual Needs (GAIN): Administration guide for the GAIN and related measures*. Bloomington, IL: Chestnut Health Systems.
- 152. Buchan, B. J., Dennis, M. L., Tims, F. M., Diamond, G. S. (2002). Cannabis use: Consistency and validity of self-report, on-site urine testing and laboratory testing. *Addiction*, *97*(1), 98-108.
- 153. Dennis, M. L., Funk, R., Godley, S. H., Godley, M. D., & Waldron, H. (2004). Cross-validation of the alcohol and cannabis use measures in the global appraisal of individual needs (GAIN) and timeline followback (TLFB; Form 90) among adolescents in substance abuse treatment. *Addiction*, 99(2), 120-128.
- 154. Dennis, M., Titus, J. C., Diamond, G., et al. (2002). The Cannabis Youth Treatment (CYT) experiment: rationale, study design and analysis plans. *Addiction*, *97*, 16-34.
- 155. Hedden, S. L., Woolson, Ř. F., & Malcolm, Ř. J. (2006). Randomization in substance abuse clinical trials. Substance Abuse Treatment and Prevention Policy, 1(6), 1-17.
- 156. Schulz, K. F., Grimes, D. A. (2002). Generation of allocation sequences in randomised trials: Chance, not choice. *The Lancet*, 359, 515-519.
- 157. Stout, R. L., Wirtz, P. W., Carbonari, J. P., Del Boca, F. K. (1994). Ensuring balanced distribution of prognostic factors in treatment outcome research. *Journal of Studies on Alcohol*, 12, 70-75.
- 158. Wei, L. J., & Lachin, J. M. (1988). Properties of the urn randomization in clinical trials. *Controlled Clinical Trials*, 9(4), 345-364.
- 159. Brown, S. A. (1989). Life events of adolescents in relation to personal and parental substance use. *American Journal of Psychiatry*, *146*, 484-489.
- 160. Dennis, M. L., Dawud-Noursi, S., Muck, R. D., & McDermeit, M. (2003). The need for developing and evaluating adolescent treatment models. In S. J. Stevens & A. R. Morral (Eds.). Adolescent drug use treatment in the United States: Exemplary models from a National Evaluation Study (3-34). Binghamton, NY: Haworth Press.
- 161. Dennis, M. L., Titus, J. C., White, M. K., Unsicker, J. I., & Hodgkins D. (2003). *Global Appraisal of Individual Needs: Administration guide for the GAIN and related measures*. Bloomington, IL: Chestnut Health Systems.
- 162. Achenbach, T. M. (1991). Integrative guide for the 1991 CBCL/4-18, YSR, and TRF profiles. Burlington, VT: University of Vermont, Department of Psychiatry.
- 163. Hudziak, J. J., Copeland, W., Stanger, C., & Wadsworth, M. (2004). Screening for DSM-IV externalizing disorders with the Child Behavior Checklist: a receiver-operating characteristic analysis. *Journal of Child Psychology and Psychiatry*, 45(7), 1299-1307.
- 164. Shelton, K. K., Frick, P. J., & Wootton, J. (1996). Assessment of parenting practices in families of elementary school-age children. *Journal of Clinical Child Psychology*, 25(3), 317-329.
- 165. McMahan, R. J., Munson, J. A., & Spieker, S. J. (1997). The Alabama Parenting Questionnaire: Reliability and validity in a high-risk longitudinal sample. Paper presented at: Association for the Advancement of Behavior Therapy. Miami, Florida.

- 166. Chapman, J.E., Sheidow A.J., Henggeler S.W., Halliday-Boykins C.A., Cunningham P.B. (2008). Developing a measure of therapist adherence to contingency management: An application of the many-facet Rasch model. *Journal of Child and Adolescent Substance Abuse*, 17(3), 47-68. PMCID: PMC2944267.
- 167. Chapman, J. E., McCart, M. R., Letourneau, E. J., & Sheidow, A. J. (2013). Comparison of youth, caregiver, therapist, trained, and treatment expert raters of therapist adherence to a substance abuse treatment protocol. *Journal of Consulting and Clinical Psychology*, 81(4), 674-680. PMCID: PMC3899684.
- 168. Pardini, D. A., Loeber, R., & Stouthamer-Loeber, M. (2005). Developmental shifts in parent and peer influences on boys' beliefs about delinquent behavior. *Journal of Research on Adolescence*, 15, 299-323.
- 169. Carver, C. S., & White, T. L. (1994). Behavioral inhibition, behavioral activation, and affective responses to impending reward and punishment: The BIS/BAS Scales. *Journal of Personality and Social Psychology*, 67(2), 319–333.
- 170. Cooper, A., Gomez, R., & Aucote H. (2007). The Behavioural Inhibition System and Behavioural Approach System (BIS/BAS) Scales: Measurement and structural invariance across adults and adolescents. *Personality and Individual Differences*, 43(2), 295–305.
- 171. Rao, H., Korczykowski, M., Pluta, J., Hoang, A., & Detre, J. A. (2008). Neural correlates of voluntary and involuntary risk taking in the human brain: an fMRI Study of the Balloon Analog Risk Task (BART). *Neuroimage*, *42*(2), 902–910.
- 172. Capaldi, D. M., & Rothbart, M. K. (1992). Development and validation of an early adolescent temperament measure. *Journal of Early Adolescence*, *12*(2), 153–173.
- 173. Ellis, L. K, & Rothbart, M. K. (2001). Revision of the Early Adolescent Temperament Questionnaire. Paper presented at: biennial meeting of the Society for Research in Child Development. Minneapolis, MN.
- 174. Casey, B. J., Trainor, R. J., Orendi, J. L., et al. (1997). A developmental functional MRI study of prefrontal activation during performance of a Go-No-Go task. *Journal of Cognitive Neuroscience*, 9, 835–847.
- 175. Davis, E. P., Bruce, J., & Gunnar, M. R. (2002). The anterior attention network: Associations with temperament and neuroendocrine activity in 6-year-old children. *Developmental Psychobiology*, 40, 43–56.
- 176. Fan, J., McCandliss, B. D., Sommer, T., Raz, A., & Posner, M. I. (2002). Testing the efficiency and independence of attentional networks. *Journal of Cognitive Neuroscience*, *14*(3), 340–347.
- 177. Higgins, S. T., Silverman, K., Heil, S. H., (Eds.) (2008). ČM in substance abuse treatment. New York, NY: Guilford.
- 178. Stanger, C., & Budney, A. J. (2010). Contingency management approaches for adolescent substance use disorders. *Child and Adolescent Psychiatric Clinics of North America*, 19(3), 547-562.
- 179. Rogers, E. M. (2003). *Diffusion of innovations*. 5th ed. New York, NY: Free Press.
- 180. Forehand, R., Lafko, N., Parent, J., & Burt, K. (2014). Is parenting the mediator of change in behavioral parent training for externalizing problems in youth? *Clinical Psychology Review*, 34, 608-619.
- 181. Blueprints for Healthy Youth Development. (n.d.). *Parent Management Training*. Retrieved from http://www.blueprintsprograms.com/factsheet/parent-management-training.
- 182. Forgatch, M. S., & Rodriguez, M. M. D. (2016). Interrupting coercion: The iterative loops among theory, science, and practice. In T. J. Dishion & J. Snyder (Eds.), *The Oxford handbook of coercive relationship dynamics* (pp. 194-214). New York: Oxford University Press.
- 183. Chamberlain P. (2003). The Oregon Multidimensional Treatment Foster Care model: Features, outcomes, and progress in dissemination. *Cognitive and Behavioral Practice*, *10*(4), 303-312.
- 184. Chamberlain, P., Price, J., Leve, L. D., Laurent, H., Landsverk, J. A., & Reid, J. B. (2008). Prevention of behavior problems for children in foster care: Outcomes and mediation effects. *Prevention Science*, 9, 17-27.
- 185. Minuchin, S. (1974). Families & family therapy. Cambridge, Mass.: Harvard University Press.
- 186. Fisher, P. A., Burraston, B., & Pears, K. (2005). The early intervention foster care program: permanent placement outcomes from a randomized trial. *Child Maltreatment*, 10(1), 61-71.
- 187 Kazdin, A. E., & Wassell, G. (2000). Therapeutic changes in children, parents, and families resulting from treatment of children with conduct problems. *Journal of the American Academy of Child and Adolescent Psychiatry*, 39(4), 414-420.

- 188. Price, J. M., Chamberlain, P., Landsverk, J., Reid, J. B., Leve, L. D., & Laurent, H. (2008). Effects of a foster parent training intervention on placement changes of children in foster care. *Child Maltreatment*, *13*(1), 64-75.
- 189. DeGarmo, D. S., Reid, J. B., Fetrow, B. A., Fisher, P. A., & Antoine, K. D. (2013). Preventing child behavior problems and substance use: The pathways home foster care reunification intervention. *Journal of Child and Adolescent Substance Abuse*, 22(5), 388-406.
- 190. Forgatch, M. S., Knutson, N. M., & Rains, L. A. (2007). A course in PMTO: The basic OSLC intervention model (Vols. 1-5). Eugene: Oregon Social Learning Center.
- 191. Patterson, G. R., & Forgatch, M. S. (1985). Therapist behavior as a determinant for client noncompliance: A paradox for the behavior modifier. *Journal of Consulting and Clinical Psychology*, 53, 846-851.
- 192. Cunningham, P. B., Randall, J., Donohue, B., & Henggeler, S. W. (2004). Contingency management supervision manual. Family Services Research Center, Medical University of South Carolina.
- 193. Sheidow, A. J., Donohue, B. C., Hill, H. H., Henggeler, S. W., & Ford, J. D. (2008). Development of an audio-tape review system for supporting adherence to an evidence-based treatment. *Professional Psychology: Research and Practice*, 39, 553-560.
- 194. Schoenwald, S. K., Sheidow, A. J., & Letourneau, E. J. (2004). Toward effective quality assurance in evidence-based practice: Links between expert consultation, therapist fidelity, and child outcomes. *Journal of Clinical Child and Adolescent Psychology*, 33, 94-104.
- 195. Schoenwald, S. K., Sheidow, A. J., Letourneau, E. J., Liao, J. G. (2003). Transportability of multisystemic therapy: Evidence for multi-level influences. *Mental Health Services Research*, 5, 223-239.
- 196. Henggeler, S. W., Schoenwald, S. K., Liao, J. G., Letourneau, E. J., & Edwards, D. L. (2002). Transporting efficacious treatments to field settings: The link between supervisory practices and therapist fidelity in MST programs. *Journal of Clinical Child and Adolescent Psychology*, 31(2), 155-167.
- 197. Muthén, L. K., & Muthén, B. O. (2015). Mplus (version 7) [computer software and manual]. Los Angeles, CA: Muthén & Muthén.
- 198. Raudenbush, S. W., & Bryk, A. S. (2002). *Hierarchical linear models: Applications and data analysis methods*. Sage Publications, Inc.
- 199. MacKinnon, D. P. (2016, April 8). Applying mediation analysis to understand how interventions work [Webinar]. In *NIH Seminar Series, Medicine: Mind the Gap*. Retrieved from https://prevention.nih.gov/programs-events/medicine-mind-the-gap/previous-seminar/applying-mediation-analysis.
- 200. MacKinnon, D. P. (2008). *Introduction to statistical mediation analysis*. New York, NJ: Lawrence Erlbaum Associates.
- 201. Singer, J. D., & Willett, J. B. (2003). *Applied longitudinal data analysis: Modeling change and event occurrence*: Oxford University Press, USA.
- 202. Cheong, J. W., MacKinnon, D. P., & Khoo, S. T. (2003). Investigation of meditational processes using parallel process latent growth curve models. *Structural Equation Modeling*, *10*, 238-262.
- 203. Biesanz, J. C., Deeb-Sossa, N., Papadakis, A. A., Bollen, K. A., & Curran, P. J. (2004). The role of coding time in estimating and interpreting growth curve models. *Psychological Methods*, 9. 30-52.
- 204. MacKinnon, D. P., Lockwood, C. M., & Williams, J. (2004). Confidence limits for the indirect effect: Distribution of the product and resampling methods. *Multivariate Behavioral Research*, 39, 99-128.
- 205. MacKinnon, D. P., Fritz, M. S., Williams, J., & Lockwood, C. M. (2007). Distribution of the product confidence limits for the indirect effect: Program PRODCLIN. *Behavior Research Methods*, 39, 384-389.
- 206. MacKinnon, D. P., Lockwood, C. M., Hoffman, J. M., West, S. G., & Sheets, V. (2002). A comparison of methods to test mediation and other intervening variable effects. *Psychological Methods*, *7*, 83-104.
- 207. Krull, J. L., & MacKinnon, D. P. (2001). Multilevel modeling of individual and group level mediated effects. *Multivariate Behavioral Research*, *36*, 249-277.
- 208. Preacher, K. J., Rucker, D. D., & Hayes, A. F. (2007). Addressing moderated mediation hypotheses: Theory, methods, and prescriptions. *Multivariate Behavioral Research*, *42*, 185-227.

- 209. Bauer, D. J., Preacher, K. J., & Gil, K. M. (2006). Conceptualizing and testing random indirect effects and moderated mediation in multilevel models: New procedures and recommendations. *Psychological Methods*, *11*, 142-163.
- 210. Cox, M. Ğ., Kisbu-Sakarya, Y., Miocevic, M., & MacKinnon, D. P. (2014). Sensitivity plots for confounder bias in the single mediator model. *Evaluation Review*, *37*, 405-431.
- 211. VanderWeele, T. J. (2010). Bias formulas for sensitivity analysis for direct and indirect effects. *Epidemiology*, *21*, 540-551.
- 212. Imai, K., Keele, L., Tingley, D. (2010). A general approach to causal mediation analysis. *Psychological Methods*, *15*, 309-334.
- 213. Mauro, R. (1990). Understanding L.O.V.E. (left out variables error): A method for estimating the effects of omitted variables. *Psychological Bulletin*, 108, 314-329.
- 214. Muthén, L. K., & Muthén, B. O. (2002). How to use a Monte Carlo study to decide on sample size and determine power. *Structural Equation Modeling*, *9*, 599-620.
- 215. Thoemmes, F., MacKinnon, D. P., & Reiser, M. R. (2010). Power analysis for complex mediational designs using Monte Carlo methods. *Structural Equation Modeling*, 17, 510-534.
- 216. Fritz, M. S., & MacKinnon, D. P. (2007). Required sample size to detect the mediated effect. *Psychological Science*, *18*, 233-239.
- 217. Nich, C., & Carroll, K. M. (2002). 'Intention-to-treat' meets 'missing data': Implications of alternate strategies for analyzing clinical trials data. *Drug and Alcohol Dependence*, *68*, 121-130.
- 218. Schafer, J. L., & Graham, J. W. (2002). Missing data: Our view of the state of the art. *Psychological Methods, 7,* 147-177.
- 219. Goldstein, H., Steele, F., Rasbash, J., & Charlton, C. (2008). REALCOM: Methodology for realistically complex multilevel modeling [computer software & manual]. Bristol, UK: Centre for Multilevel Modelling.
- 220. Molenberghs, G. & Verbeke, G., (2006). Models for discrete longitudinal data. New York: Springer.
- 221. Hedeker, D., & Gibbons, R. D. (1997). Application of random-effects pattern-mixture models for missing data in longitudinal studies. *Psychological Methods*, 2, 64-78.